CLINICAL TRIAL: NCT05998824
Title: COVID-19 Vaccination Hesitancy in Adults With Sickle Cell Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: American Society of Hematology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00110966
Record Dates: First submitted 2023-08-17; First posted 2023-08-21 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-06

CONDITIONS: Sickle Cell Disease; COVID-19 Vaccine; Vaccine Hesitancy
MeSH Terms: conditions — Anemia, Sickle Cell; Vaccination Hesitancy | interventions — Videotape Recording

STUDY DESIGN:
Intervention Model Description: measurement by survey before and after intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adults With Sickle Cell Disease (Other): Age 18 years or older
  Interventions: Behavioral: SCD-specific COVID-19 vaccination information (SCVI) video

INTERVENTIONS:
Behavioral: SCD-specific COVID-19 vaccination information (SCVI) video — SCD-specific COVID-19 vaccination information (SCVI) video developed by health care providers with input from a community advisory board of people with sickle cel disease and their caregivers.
  Other Names: Video

SUMMARY:
The goal of this clinical trial is to test an COVID-19 vaccination information video in adults with sickle cell disease. The main questions it aims to answer are why are some adults with sickle cell disease hesitant to receive COVID-19 vaccination and whether a COVID-19 vaccination information video tailored for people with sickle cell disease will reduce vaccine hesitancy. Participants will complete a brief survey before and after watching a short video with information on vaccine safety, efficacy, and the greater impact of COVID-19 infection on people with sickle cell disease.

DETAILED DESCRIPTION:
In this research study, we seek to gain a better understanding of reasons for COVID-19 vaccine hesitancy in adults with sickle cell disease (SCD). We will develop a SCD-specific COVID-19 vaccination information (SCVI) video that discusses vaccine safety, efficacy, and necessity of COVID-19 vaccination for the sickle cell patient population, and determine if the video reduces vaccine hesitancy in adults with SCD. Hopefully, this will inform future education interventions to improve confidence in COVID-19 vaccines and subsequently increase vaccination rates.

Specifically, the research objectives are:

To determine factors associated with COVID-19 vaccine hesitancy in adults with SCD To determine if a SCD-specific COVID-19 vaccination information (SCVI) video reduces vaccine hesitancy in adults with SCD.

This study will be conducted as a part of an ongoing prospective research study aimed at better understanding COVID-19 vaccine hesitancy at the Duke Adult Comprehensive Sickle Cell Center. Two cross-sectional surveys will be administered to patients seen in the Adult Sickle Cell Clinic and Day Hospital who meet the inclusion criteria. The purpose of the initial survey will be to obtain a baseline vaccination rate and to gain a better understanding behind vaccine hesitancy in this patient population. After completion of the first survey, a short video discussing the safety, efficacy, and importance of the COVID-19 vaccine for patients with sickle cell disease will be watched prior to completing the second survey. The video will be available via scanning a QR code or via direct link if the survey is filled out electronically. Members of the Community Advisory Board for the Duke Sickle Cell Program will be interviewed in a group to gain an understanding of how to improve and implement the assessment in practice (non-research activity). A subsequent "post-intervention" survey will then administered to determine if the SCVI video reduces vaccine hesitancy in adults with SCD. Both surveys should take ~5 minutes to complete. We estimate that these surveys will reach ~250 patients over the six months they are administered. Informed consent will obtained prior to completion of the surveys and watching the video. Survey responses will remain anonymous with no patient identifying information required for completion. Data will be stored and protected using the secure REDCap database.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of sickle cell disease

Exclusion Criteria:

* unable to read or understand spoken English to complete the survey

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 33 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Vaccine hesitancy | before and after watching video
  To assess vaccine hesitancy in patients not vaccinated for COVID-19, we will ask participants "how likely are you to get vaccinated for COVID-19 in the future?". Response options will be dichotomized into not hesitant ("likely or somewhat likely") vs neutral vs hesitant ("somewhat unlikely or not likely"). We will also assess vaccine hesitancy for people

CONTACTS AND LOCATIONS:
Overall Officials: John Strouse, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Adult Sickle Cell Program, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No